CLINICAL TRIAL: NCT05602584
Title: The Effect of Immunophenotype on Prognosis of Sepsis
Brief Title: Effect of Immunophenotype on Prognosis of Sepsis
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jianfeng Xie, Clinical Professor, Southeast University, China
Other Study IDs: EOIPOPOS
Record Dates: First submitted 2022-07-02; First posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Sepsis; Septic Shock; Sepsis Syndrome
Keywords: Immunophenotype
MeSH Terms: conditions — Sepsis; Shock, Septic; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — Peripheral blood of patients with sepsis was collected on day 1, 3, 7, 14 and 28
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The popuse of this study is to assess the inflammatory immunophenotypes of sepsis patients are significantly correlated with prognosis, which may provide theoretical basis for precise immune regulation of sepsis.

DETAILED DESCRIPTION:
The clinical characteristics and inflammatory/immune markers of sepsis patients were analyzed dynamically and followed up to one year after diagnosis. Through latent category analysis, cluster analysis and other inflammatory immunophenotypes, the clinical characteristics of different inflammatory immunophenotypes and their relationship with the long-term prognosis of sepsis were clarified.

ELIGIBILITY:
Inclusion Criteria:Patients with sepsis 3 diagnostic criteria were admitted to ICU; Aged 18 or above; Within 24 hours of diagnosis.

-

Exclusion Criteria:Malignant tumor; Autoimmune diseases; Diseases of the blood system; HIV infection; History of high-dose glucocorticoid use (hydrocortisone 200mg/d or other hormone with equivalent titer, more than one week); pregnancy

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We investigate the patients with sepsis 3 diagnostic criteria were admitted to ICU; Aged 18 or above; Within 24 hours of diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
survival or death in 28 days | From date of randomization until the date of out of ICU or date of death from any cause, whichever came first, assessed up to 28 days
  observe wether the patients is survival or death in 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Critical Care , Zhong-da Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No